CLINICAL TRIAL: NCT04168632
Title: Fostering Sustainable Dietary Habits Through Optimized School Meals - an Intervention Study
Brief Title: Fostering Healthy and Sustainable Diets Through School Meals
Acronym: OPTIMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Göteborg University (Other); University College Copenhagen (Other)
Responsible Party: Principal Investigator, Liselotte Schäfer Elinder, professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-00353; 2016-00353 (Other Grant/Funding Number: Formas)
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Food Habits
Keywords: children; public meals; sustainable diets; Agenda 2030
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Three schools from one municipality in the Region Stockholm met inclusion criteria and were eligible to participate in the intervention. These schools all served the baseline followed by the new menu. Each period lasted four weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A new 4-week menu plan
  Interventions: Other: OPTIMAT

INTERVENTIONS:
Other: OPTIMAT — The intervention was to serve a new school lunch menu plan as similar as possible to a baseline menu plan but 40% lower in greenhouse gas emissions, being nutritionally adequate and no more expensive.

SUMMARY:
School meals have considerable potential to shape children's diets and reduce the climate impact of meals. This study applies linear programming for developing and implementing a climate friendly, nutritious and affordable school lunch menu. The new menu plan will be compared to the baseine menu during a 4-week intervention trial. The outcomes will be food waste, consumption, and pupils' satisfaction with the meals before and after introducing the new meal plan by interrupted time series analysis. Our hypothesis is that school meals can be optimized to be nutritious and more climate friendly, without negatively affecting acceptance, food waste and cost.

A number of primary schools in one Swedish municipality with the same menu plan for all schools participated in the study. Their current meal supply was recorded in the form of a food list including amount and cost of each item over a 4-week period. This list was then optimized with linear programming to be as similar as possible to the baseline diet but with a 40% reduction in greenhouse gas emissions. No new foods were introduced and none were removed from the list. Nutritionally adequacy was ensured by included constraints into the model. The optimized food list was handed to a professional meal planner and a new menu plan was developed based on the revised food list. Data on food waste and consumption was collected daily during a baseline period of four weeks, and during the four-week intervention period. School lunch satisfaction was assessed twice with an online questionnaire at baseline and during the intervention. After the end of intervention, students and meal staff were interviewed regarding their experiences with the new meals.

DETAILED DESCRIPTION:
For a period of four weeks, during the spring term of 2019, Swedish primary school children received a new school lunch menu plan which was optimized through linear programming to be as similar to the baseline menu as possible with 40% lower in greenhouse gas emissions (GHGE), is nutritionally adequate, and not more expensive.

Primary schools in three municipalities in the Stockholm Region were invited to the trial via their chief meal strategist. To be included in the intervention, the schools had to have in-house food preparation (i.e. not serve catered food) and be able to provide recipes for a standard four-week menu plan electronically (critical for the optimization process). Three schools from one of the municipalities met inclusion criteria and were thus eligible to participate in the intervention.

Recipes for an original (baseline) four-week school lunch menu plan previously served at the recruited schools were obtained through the municipality's electronic meal planning system. Each food item included has a code that can be coupled to the national food database and a national climate database for foods (Research Institutes of Sweden). These foods were considered as the baseline food supply needed to compose a new four-week school lunch menu plan. The list of foods and amounts was optimized using linear programming to be as similar as possible to the baseline list. The optimized food list was then handed to a professional meal planner who developed a new menu plan for the intervention, using all foods in the optimized food list.

To assess the effect of the new menu plan, data on daily food waste and consumption was collected at school level in each intervention school four weeks before (baseline) as well as during the four-week intervention period with a 2-week brake between measurement periods. A tool for measuring food waste and consumption in school restaurants developed by the National Food Agency in Sweden was used. The tool required weighting of all kitchen waste (both preparation waste and cooking waste); all food prepared in the kitchen; the share of the prepared food that was served but not eaten by the pupils and had to be thrown away (serving waste); the share that could be saved for future meals; and plate waste. The daily number of plates used by the pupils in the school restaurant was also recorded. These measurements were made daily by the personnel in the school kitchens during baseline as well as during the intervention period.

Data on school meal satisfaction was measured through an online questionnaire at baseline and during the last week of the intervention. Pupils in grades 5 and 8 answered the questionnaire that contained ten questions related to the school lunch. Five of the ten multiple-choice questions specifically covered their general (i.e. not for that specific day of week) sense of satisfaction with the school lunch.

Six focus group discussions (FGD) with pupils in grades 5 and 8 and three FGDs with meal staff will be conducted to explore their experiences with the intervention as well as the barriers and facilitators to scaling up.

ELIGIBILITY:
Inclusion Criteria:

* Primary schools (year 0-9)
* The schools needed to have on-site kitchens
* The schools needed to be able to provide previously used recipes for a standard four-week menu electronically

Exclusion Criteria:

* Preschools or gymnasiums
* Schools receiving catered food
* Schools that could not provide recipes electronically

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1635 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in food waste between baseline and intervention periods | During four weeks before the intervention period and during the four week intervention.
  Kitchen waste, serving waste, and plate waste, total per school and per pupil
Change in food consumption between baseline and intervention periods | During four weeks before the intervention period and during the four week intervention.
  Food consumption, total per school and per pupil
Change in school meal satisfaction between baseline and intervention periods | Once during the four weeks preceding the intervention as well as once during the last week of intervention.
  Pupils' rating of school meals with the "SkolmatSverige" student questionnaire (ten questions referring to the school lunch with face validity with a varying number of response options)

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte Schäfer Elinder, professor, Principal Investigator — Karolinsk Institutet
Locations (1):
- Botkyrka municipality, Stockholm, Botkyrka, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eustachio Colombo P, Patterson E, Schafer Elinder L, Lindroos AK, Sonesson U, Darmon N, Parlesak A. Optimizing School Food Supply: Integrating Environmental, Health, Economic, and Cultural Dimensions of Diet Sustainability with Linear Programming. Int J Environ Res Public Health. 2019 Aug 21;16(17):3019. doi: 10.3390/ijerph16173019. PMID 31438517
- [Derived] Eustachio Colombo P, Elinder LS, Patterson E, Parlesak A, Lindroos AK, Andermo S. Barriers and facilitators to successful implementation of sustainable school meals: a qualitative study of the OPTIMAT-intervention. Int J Behav Nutr Phys Act. 2021 Jul 3;18(1):89. doi: 10.1186/s12966-021-01158-z. PMID 34217304
- [Derived] Eustachio Colombo P, Patterson E, Lindroos AK, Parlesak A, Elinder LS. Sustainable and acceptable school meals through optimization analysis: an intervention study. Nutr J. 2020 Jun 24;19(1):61. doi: 10.1186/s12937-020-00579-z. PMID 32580743

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/32/NCT04168632/Prot_SAP_000.pdf